CLINICAL TRIAL: NCT03043157
Title: Rocuronium ED50 for Excellent Laparoscopic Conditions for Cholecistectomy: Dose-finding Adaptative Clinical Trial
Brief Title: Rocuronium Effective Dose for Laparoscopic Cholecystectomy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Brasilia University Hospital (Other)
Responsible Party: Principal Investigator, Gabriel Magalhaes Nunes Guimaraes, Head of Anesthesiology, Brasilia University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CAAE 60322116.2.0000.0025
Record Dates: First submitted 2017-02-02; First posted 2017-02-03 (Estimated); Last update posted 2017-09-13 (Actual); Status verified 2017-09

CONDITIONS: Muscle Relaxation
MeSH Terms: interventions — Rocuronium

STUDY DESIGN:
Intervention Model Description: Dose-finding using Dixon's up-and-down adaptative clinical trial
Masking Description: Participant receives hypnotic (propofol) before we use the drug
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dose-finding group (Other): The first patient will receive rocuronium 0,6mg/kg. After that, every patient's dose will depend on the outcome of the previous patient. It will go up 0,1mg/kg if the laparoscopic conditions were not excellent or go down 0,1mg/kg otherwise.
  Interventions: Drug: rocuronium

INTERVENTIONS:
Drug: rocuronium — intravenous rocuronium infusion

SUMMARY:
This is an adaptative study where each participant's rocuronium dose will depend on the previous patient's response, being higher if it was not enough and lower if it was more than enough.

DETAILED DESCRIPTION:
Rocuronium is one of the most used neuromuscular blockers to help intubation and to relax abdominal wall for laparoscopic surgery.

Rocuronium intubation dose can be enough for intubation but not last enough for excellent laparoscopic conditions. There is little variation in time from anesthesia induction to the end of the laparoscopy for cholecystectomy and avoiding excess rocuronium dose can help providing excellent conditions and fast track extubation.

Dixon's up-and-down method will guide this dose-finding study for the ED50.

ELIGIBILITY:
Inclusion Criteria:

* general anesthesia

Exclusion Criteria:

* deny participation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2017-02-15 (Actual); Primary Completion 2017-03-02 (Actual); Study Completion 2017-03-02 (Actual)

PRIMARY OUTCOMES:
Excellent laparoscopic conditions | 30 minutes
  Subjective laparoscopic conditions for surgery, assessed by the main surgeon, as excellent or not

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel MN Guimaraes, MsC, Principal Investigator — Universidade de Brasilia
Locations (1):
- Hospital das Forças armadas, Brasília, Federal District, Brazil

IPD SHARING:
Plan to Share IPD: No